CLINICAL TRIAL: NCT04847739
Title: Seeded Cells on Matrix Plug Treating Crohn's Perianal Fistulas (STOMP-II)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Avobis Bio, LLC (Industry)
Collaborators: Alimentiv Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STOMP-II
Record Dates: First submitted 2021-04-01; First posted 2021-04-19 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Perianal Fistula; Crohn's Disease
Keywords: Matrix plug; Mesenchymal stem cells; Fistula plug; Refractory; Recurrent; STOMP; Autologous
MeSH Terms: conditions — Crohn Disease; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care Treatment + AVB-114 (Experimental): Subjects receive the standard of care treatment (seton placement) prior to Day 0, when it is removed and the AVB-114 study treatment is inserted.
  Interventions: Procedure: Seton Placement; Drug: AVB-114
- Standard of Care Treatment (Active Comparator): Subjects receive the standard of care treatment (seton placement) prior to Day 0, when it is removed and then replaced.
  Interventions: Procedure: Seton Placement

INTERVENTIONS:
Procedure: Seton Placement — This treatment consists of inserting a seton (a soft flexible tube or nonabsorbable string) into the subject's perianal fistula. The seton will be removed by a study doctor at study visits as applicable.
Drug: AVB-114 — AVB-114 consists of stem cells taken from a subject's fat tissue seeded into a bioabsorbable plug. AVB-114 will be inserted into the subject's fistula by a study doctor on Day 0.
  Arms: Standard of Care Treatment + AVB-114

SUMMARY:
A Phase II study to assess the safety and efficacy of AVB-114 in treatment of complex Crohn's perianal fistulas in subjects with quiescent rectal disease and whose fistula has failed to respond to biologic or conventional therapy. Combined remission of treated perianal fistula in the investigational treatment arm will be compared to a standard of care control arm.

The study has 2 parts:

Part 1: All required study visits for subjects who initially receive study treatment and those who receive standard of care therapy (control arm).

Part 2: Subjects who are enrolled in the control arm may receive treatment with AVB-114 following week 36. Those subjects then will be followed as specified in the clinical protocol.

DETAILED DESCRIPTION:
AVB-114 is an investigational therapy which offers a new therapeutic approach to treating this unmet medical need. The drug product is a mesenchymal cell substrate system comprised of autologous mesenchymal cells incubated with a 3-dimensional bioabsorbable substrate. The drug substance is expanded, pure mesenchymal stem cells (MSC) which are known to modulate local inflammation and orchestrate tissue healing. By incubating cells with a 3-dimensional bioabsorbable substrate designed for anal fistula geometry, cells are locally delivered into the fistula tract to promote healing.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated ICF.
2. Ability and willingness to comply with study protocol and study requirements for the duration of the study.
3. Male or female, 18-70 years of age
4. Subjects with CD diagnosed at least 6 months prior to screening visit.
5. Subjects with a single fistula tract with one internal opening and one external opening.
6. Subjects whose perianal fistula(s) were previously treated with either biologic or conventional therapy whose fistula has demonstrated a failed response or who have documented medication intolerance.
7. Women of childbearing potential (WCBP) must have negative serum pregnancy test at screening (sensitive to 25 IU human chorionic gonadotropin). WCBP participating in this study must agree to use an adequate method of contraception during the entire duration of the study. Males who have sexual partners that are women of childbearing potential must be willing to use a barrier method for contraception for the duration of study.

Exclusion Criteria:

1. Clinically significant medical conditions within the six months before screening that would, in the opinion of the investigator, compromise the safety of the subject with study participation and/or the ability of the subject to follow study protocol.
2. Evidence of hepatitis B, C, or HIV or subjects with congenital or acquired immunodeficiencies.
3. Participation in an investigational drug study (within 30 days of last administration from screening visit) or investigational medical device study (within 1 year of implant from screening visit) where investigational treatment (drug or device) is placed in rectum, vagina, or near fistula location, or that may potentially interact with study treatment.
4. History (within previous 5 years of screening visit) of invasive cancer including melanoma (with the exception of localized skin cancers).
5. Subjects pregnant, trying to become pregnant, or are breast feeding.
6. Subjects with known allergies or hypersensitivity to aminoglycosides and contraindications to Magnetic Resonance (MR) evaluations and/or to MR contrast.
7. History of clinically significant fat-directed autoimmunity.
8. Genito-urinary fistulization, including rectovaginal (i.e., fistulae that transverse the vaginal canal).
9. Presence of an ileal anal pouch.
10. Active, unresolved infection requiring parenteral antibiotics.
11. Any major surgery of the gastrointestinal tract (including one or more segments of the colon or terminal ileum) within 3 months prior to screening visit. Presence of stoma is not exclusionary.
12. Subjects who had a definitive surgical procedure for the target fistula or a perianal procedure that resulted in a large soft tissue defect within 6 months prior to screening visit.
13. Subjects where the target adipose collection harvest site is compromised due to a previous cool sculpting procedure, local radiation, chemotherapy, recent tattoos, local infection, or other reasons that may compromise the adipose tissue for study use.
14. Subjects previously treated with Cx601/Alofisel or other allogeneic or autologous stem-cell therapy within the past 6 months.
15. Contraindications to the anesthetic procedure (local and general) or to the adipose tissue collection procedure.
16. Subjects with one or more of the following fistula types or anatomic presentations:

    1. Horseshoe fistulas
    2. Fistulas that do not have an opening inside the anal canal or low rectum
    3. Blind ending sinus tracts (no external opening)
    4. Branching fistulas. A previously performed conversion of a branching fistula tract to a single tract is not exclusionary
    5. >1 internal opening
    6. Moderate or severe proctitis
    7. Severe rectal mucosal fibrosis surrounding the internal opening preventing the securing of the fistula plug cap.
    8. Any anatomical limitation to successfully securing the fistula plug cap
17. Evidence by colonoscopy of moderately or greater active luminal CD.
18. Subject with ongoing systemic or rectal steroids for CD in the last 2 weeks prior to screening and baseline study visits.
19. History of, or concurrent high-grade dysplasia, adenocarcinoma, and carcinoma in situ on colonoscopy within 5 years of screening visit.
20. Subjects with renal insufficiency (creatinine value > 1.8 mg/dL, eGFR < 44, or patient undergoing dialysis).
21. Subjects with a hemoglobin less than 8 gm/dL.
22. Subjects with serum aspartate transaminase (AST) or alanine transaminase (ALT) > 2 times the upper limit of normal (ULN).
23. Subjects with an abscess within the fistula tract that cannot be resolved prior to treatment.
24. Subjects with known coagulopathy (abnormal INR) or thrombocytopenia as indicated by a platelet count < 75,000.
25. Subjects with history of substance abuse (drug or alcohol) that would interfere with the ability to comply with the study protocol and study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in proportions of subjects with combined remission of treated perianal fistula between the AVB-114 and standard of care groups. | 36 weeks

SECONDARY OUTCOMES:
Change in proportions of subjects with fistula clinical remission between the AVB-114 and standard of care groups. | Week 12 to Week 104
Change in the means of durability of clinical remission between the AVB-114 and standard of care groups. | Week 12 to Week 104
  Length of time fistula meets clinical remission definition.
Change in means of time to clinical remission between the AVB-114 and standard of care groups. | Week 12 to Week 104
Change in proportions of subjects with fistula relapse between the AVB-114 and standard of care groups. | Week 12 to Week 104
Change in means of time to fistula relapse between the AVB-114 and standard of care groups. | Week 12 to Week 104
Change in proportions of radiologic response of treated fistula between the AVB-114 and standard of care groups. | Baseline, Week 12 to Week 52
Change in means of disease activity index scores using the Perianal Disease Activity Index (PDAI) between the AVB-114 and standard of care groups. | Baseline, Week 36
  Perianal Disease Activity Index (PDAI). Possible scores range from 0-20, with a higher score indicating more severe perianal disease activity
Change in means of disease activity index scores using the short Crohn's Disease Activity Index (sCDAI) between the AVB-114 and standard of care groups. | Baseline, Week 36
  Short Crohn's Disease Activity Index (sCDAI). Possible scores range from 44 to >450, with a higher score representing more severe disease activity
Change in means of patient quality of life assessment scores using the Euroqol 5 Diumention 5, level measure of health status (Eq-5Q-5L) between the AVB-114 and standard of care groups. | Baseline, Week 36
  Euroqol 5 Dimension 5, level measure of health status (EQ-5D-5L). The scale ranges in scores from 0 to 100, with a higher score indicating a more severe health status.
Change in means of patient quality of life assessment scores using the Inflammatory Bowel Disease Questionnaire (IBDQ) between the AVB-114 and standard of care groups. | Baseline, Week 36
  Inflammatory Bowel Disease Questionnaire (IBDQ). Possible scores range from 32-224, with a higher score indicating a better health-related quality of life.
Change in patient assessment of impact to daily functionality related to treated fistula between the AVB-114 and standard of care groups. | Baseline, Week 12 to Week 36
  Days of missed work or activity and reason why will be captured.
Change in the evaluations of patient care trajectory related to treated fistula between the AVB-114 and standard of care groups. | Week 12 to Week 36
  Number and type of healthcare resources utilized will be captured.
Change in number of adverse events between the AVB-114 and standard of care groups. | Day 1 to Week 104
Change in number of serious adverse events between the AVB-114 and standard of care groups. | Day 1 to Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Joan Morris, Study Director — Alimentiv Inc.
Locations (15):
- United States (15):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Office of Phillip Fleshner, MD, Los Angeles, California
  - Stanford University, Redwood City, California
  - UC Davis, Sacramento, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - UChicago Medicine and Biological Sciences, Chicago, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Mass Gen Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical College - NY Presbyterian Hospital, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No